CLINICAL TRIAL: NCT01107496
Title: A Phase I/IIa Randomized, Double-Blind, Multicenter, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Immediate-Release Viloxazine in Adults With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: Evaluation of Immediate-Release Viloxazine in Adults With ADHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 812P201
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Attention-Deficit/Hyperactivity Disorder (ADHD)
Keywords: ADHD; Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IR Viloxazine (Experimental): Treatment A: immediate-release (IR) viloxazine capsules administered orally 3 times a day
  Interventions: Drug: IR Viloxazine
- Placebo (Placebo Comparator): Treatment B: Placebo capsules administered orally 3 times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IR Viloxazine — One 50mg immediate-release viloxazine capsule administered orally 3 times a day (150mg total daily dose) for Week 1.
  Two 50mg immediate-release viloxazine capsules administered orally 3 times a day (300mg total daily dose) for Weeks 2 to 6.
  Other Names: immediate-release viloxazine; SPN-812V immediate-release
  Arms: IR Viloxazine
Drug: Placebo — Placebo capsules administered orally 3 times a day
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, parallel group, safety and tolerability study in adults with ADHD. The target subjects are healthy male or female adults aged 18 to 64 years, inclusive, with a diagnosis of ADHD.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, multicenter, placebo-controlled, parallel group, safety and tolerability study in adults with ADHD. The target subjects are healthy male or female adults aged 18 to 64 years of age, inclusive, with a diagnosis of ADHD. Approximately 50 subjects will be enrolled at approximately 5 sites in the United States. Subjects will be randomized (1:1) to one of two treatment groups, immediate-release (IR) viloxazine or placebo. Primary objective is to determine the safety of IR viloxazine in adults with ADHD.

ELIGIBILITY:
Inclusion criteria:

1. Able to provide informed consent prior to any study procedure being conducted.
2. Capable and willing to comply with study procedures.
3. Male or female aged 18 to 64, inclusive.
4. Subjects with a current diagnosis of ADHD as confirmed by the Conners' Adult ADHD Diagnostic Interview for DSM-IV (CAADID)
5. Clinical Global Impression - Severity (CGI-S) score of 4 or higher.
6. On no treatment for ADHD or willing to be withdrawn from an ongoing treatment after a washout of at least 10 days.
7. Body Mass Index (BMI) between 18.0 and 34.0 inclusive.
8. Subject must be in general good health as determined by medical history, ECG, and other analysis that, in the judgment of the Investigator, would confirm the Subject's good health.
9. Females of childbearing potential (FOCP) who, if sexually active, agree to use acceptable forms of contraception (including oral, transdermal, or implanted contraceptives; intrauterine device; female condom with spermicide; diaphragm with spermicide; cervical cap; abstinence; use of condom with spermicide by sexual partner or sterile [at least 6 months prior to SM administration] sexual partner) at least 14 days prior to start of study drug administration, throughout the study, and for 30 days following the last dose of SM.
10. Postmenopausal females with amenorrhea for at least 2 years or females who are permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy).

Exclusion Criteria

1. Current or past history of psychotic disorder or major depressive disorder with psychotic features.
2. Presence of another primary DSM-IV-TR disorder.
3. Suicidality, defined as either active suicidal plan/intent or active suicidal thoughts, in the 6 months before the Screening Visit or more than 1 lifetime suicide attempt. (The Columbia-Suicide Severity Rating Scales [C-SSRS] will be administered at each visit.)
4. Substance or alcohol abuse/dependence within previous 6 months, or a positive urine drug screen at screening or baseline prior to first dose of study medication (SM).
5. Any known or suspected significant medical or psychiatric illnesses that, in the judgment of the Investigator, may impair interpretation of study results or constitute a significant safety concern in the context of the clinical trial
6. ECG abnormalities (clinically significant according to Investigator's opinion) or vital sign abnormalities (systolic blood pressure [SBP] <90 or >140 millimeters of mercury [mmHg], diastolic blood pressure [DBP] <40 or >90mmHg, or heart rate [HR] <40 or >100 beats per minute [BPM]) at screening.
7. Clinically significant laboratory abnormalities; including presence of potential hepatic function impairment as shown by, but not limited to alanine aminotransferase (ALT/SGPT) values >2 times upper limit of normal (ULN), aspartate aminotransferase (AST/SGOT) > 2 times ULN, gamma-glutamyl transpeptidase (GGT) >3 times ULN, or total bilirubin >1.5 ULN .
8. Medications, including health food supplements judged by the Investigator to be likely to have central nervous system activity (for example, St John's Wort, gingko leaf, and melatonin), are not permitted during the study. If the subject is taking the medication prior to study entry, there must be a 7 day washout period prior to first dose of SM.
9. Lifetime history of tic disorder, Tourette's Disease, or organic brain disorder; or family history of Tourette's Disease.
10. Current or lifetime history of hyperthyroidism unless treated and stable for at least 6 months.
11. Participation in or plan to begin behavioral therapy during the study.
12. Subject has a prior history of allergy or any significant adverse reaction (including rash) to study medication, or any of the product components.
13. Females who are pregnant or lactating or are unwilling to use an acceptable form of contraception throughout the study.
14. Difficulty swallowing whole capsules.
15. History of seizures or risk factors for seizures (e.g., head trauma), not including febrile seizures.
16. Use of an investigational drug or participation in an investigational study within 30 days prior to first dose of SM.
17. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Rubin, MD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (4):
- United States (4):
  - Bradenton, Florida
  - Libertyville, Illinois
  - Owensboro, Kentucky
  - Herndon, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Treatment B: Placebo administered orally 3 times a day
Period: Overall Study
Arm/Group | IR Viloxazine | Placebo
Started (Subjects who were randomly assigned to one of two treatment groups (Randomized Population).) | 26 | 26
Dosed (Subjects who were randomly assigned to one of two treatment groups and took at least one dose of study medication (Safety Population)) | 26 | 25
Completed | 24 | 24
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population, defined as subjects who were randomly assigned to one of two treatment groups and took at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | IR Viloxazine | Placebo | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.7 (14.04) | 43.1 (10.39) | 40.4 (12.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 12 | 16 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 24 | 48
  Asian | 0 | 1 | 1
  Other | 2 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 25 | 25 | 50
Height [Mean (Standard Deviation); unit: inches] | 66.740 (3.5103) | 68.406 (4.0851) | 67.557 (3.8573)
Weight [Mean (Standard Deviation); unit: pounds (lbs)] | 163.85 (33.641) | 171.05 (33.057) | 167.38 (33.221)
BMI [Mean (Standard Deviation); unit: kilograms per square meter] | 25.688 (3.7216) | 25.664 (4.3620) | 25.676 (4.0073)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events During 6 Weeks of Treatment
Description: The percent of subjects who took at least one dose of immediate-release viloxazine (Safety Population; N) and who reported at least one Adverse Event (n). The percent is calculated by dividing "the number of subjects who reported at least one Adverse Event (n)" by "the number of subjects in the Safety Population (N)" and multiplying the product by 100. The higher the percentage, the higher the incidence in the Safety Population
Time Frame: Weeks 1-6
Population: Safety Population (N), defined as subjects who were randomly assigned to one of two treatment groups and took at least one dose of study medication.
Measure: Number; unit: percentage of subjects
Arm/Group | IR Viloxazine | Placebo
Number analyzed (Participants) | 26 | 25
percentage of subjects | 88.5 | 72.0

2. Secondary Outcome: Change From Baseline in the Investigator-Rated Conners' Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale (CAARS) Total Score at Week 6 (End of Study)
Description: The Conners' Adult ADHD Rating Scale (CAARS) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology in adults. The CAARS consists of 30 items, including 18 items that correspond to the 18 ADHD symptoms per the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV). The 18 items are further subdivided into two subscales: Inattention (9 items) and Hyperactivity/Impulsivity (9 items). Each item is rated on a 4-point scale from 0 (not at all, never) to 3 (very much, very frequently). The sum of 18 items yields the raw Total score (range: 0 to 54; the higher the score, the more severe the ADHD symptoms). Raw score is converted to a change from baseline (CFB) score. A lower CFB score (<0) represents a better outcome.
Time Frame: Baseline and Week 6
Population: Intent-to-Treat (ITT) Population (N), defined as subjects who were randomly assigned to one of two treatment groups, took at least one dose of study medication, had a valid baseline CAARS assessment (pre-dosing), and had at least one valid post-baseline CAARS assessment.
Measure: Median (Full Range); unit: units on a scale
Groups:
- IR Viloxazine: Immediate-release (IR) viloxazine capsules administered orally 3 times a day
- Placebo: Placebo administered orally 3 times a day
Arm/Group | IR Viloxazine | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale
  Raw score; Baseline | 36.0 [20 to 54] | 35.0 [21 to 45]
  Change from Baseline score; Week 6 | -11.5 [-38 to 4] | -6.0 [-34 to 6]
Statistical Analysis 1: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 6 data; Test type: Superiority; p = 0.0414, Wilcoxon (Mann-Whitney); Median Difference (Net) = 6.00, 95% CI 2-sided [1.00 to 12.00]

3. Secondary Outcome: Change From Baseline in the Investigator-Rated Conners' Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale (CAARS) Total Score at Week 1
Description: as for outcome 2
Time Frame: Baseline and Week 1
Population: Intent-to-Treat (ITT) Population (N), defined as subjects who were randomly assigned to one of two treatment groups, took at least 1 dose of study medication, had a valid baseline CAARS assessment (pre-dosing), and had at least one valid post-baseline CAARS assessment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IR Viloxazine | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale
  Raw score; Baseline | 36.0 [20 to 54] | 35.0 [21 to 45]
  Change from Baseline score; Week 1 | -5.0 [-29 to 1] | -2.0 [-25 to 7]
Statistical Analysis 1: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 1 data; Test type: Superiority; p = 0.0803, Wilcoxon (Mann-Whitney); Median Difference (Net) = 3.00, 95% CI 2-sided [0.00 to 7.00]

4. Secondary Outcome: Change in Global Clinical Impression-Improvement (CGI-I) Score From Baseline Global Clinical Impression-Severity of Illness (CGI-S) Score at Week 1, Week 2, Week 3, Week 4, Week 5, and Week 6
Description: The Global Clinical Impression-Improvement (CGI-I) scale is a single item clinician-rated assessment of how much the subject's condition (symptoms) has improved, worsened, or has not changed relative to his/her baseline state prior to the beginning of treatment; it is rated on a 7-point scale from 1 to 7, where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. The Clinical Global Impression-Severity of Illness (CGI-S) score is a single item clinician-rated assessment of the severity of subject's condition (symptoms) in relation to the clinician's total experience with patients with ADHD; it is rated on a 7-point scale with 1=Normal, not at all ill, 2=Borderline Ill, 3=Mildly Ill, 4=Moderately Ill, 5=Markedly Ill, 6=Severely Ill, 7=Among the most extremely ill patients. CGI-I scores at post-baseline visits were subtracted from CGI-S score at baseline; a change from baseline score <0 represent better outcome.
Time Frame: Weeks 1, 2, 3, 4, 5, and 6
Population: Intent-to-Treat (ITT) Population (N), defined as subjects who were randomly assigned to one of two treatment groups, took at least 1 dose of study medication, had a valid CGI-S assessment at baseline, and had at least one valid post-baseline CGI-I assessment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IR Viloxazine | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale
  Change from "Baseline CGI-S Score"; Week 1 | 0.0 [-2 to 5] | 0.0 [-1 to 4]
  Change from "Baseline CGI-S Score"; Week 2 | -1.0 [-2 to 5] | 0.0 [-2 to 4]
  Change from "Baseline CGI-S Score"; Week 3 | -1.5 [-2 to 4] | 0.0 [-2 to 4]
  Change from "Baseline CGI-S Score"; Week 4 | -1.5 [-3 to 4] | 0.0 [-2 to 5]
  Change from "Baseline CGI-S Score"; Week 5 | -1.5 [-3 to 4] | 0.0 [-2 to 4]
  Change from "Baseline CGI-S Score"; Week 6 | -1.0 [-3 to 4] | 0.0 [-1 to 4]
Statistical Analysis 1: Comparison: IR Viloxazine; This analysis pertains to Week 1 data; Test type: Superiority; p = 0.5308, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.00, 95% CI 2-sided [-1.00 to 1.00]
Statistical Analysis 2: Comparison: IR Viloxazine vs Placebo; This analysis pertains to Week 2 data; Test type: Superiority; p = 0.2032, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.00, 95% CI 2-sided [-2.00 to 0.00]
Statistical Analysis 3: Comparison: IR Viloxazine vs Placebo; This analysis pertains to Week 3 data; Test type: Superiority; p = 0.0677, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.00, 95% CI 2-sided [-2.00 to 0.00]
Statistical Analysis 4: Comparison: IR Viloxazine vs Placebo; This analysis pertains to Week 4 data; Test type: Superiority; p = 0.0743, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.00, 95% CI 2-sided [-2.00 to 0.00]
Statistical Analysis 5: Comparison: IR Viloxazine vs Placebo; This analysis pertains to Week 5 data; Test type: Superiority; p = 0.0437, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.00, 95% CI 2-sided [-2.00 to 0.00]
Statistical Analysis 6: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 6 data; Test type: Superiority; p = 0.1209, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.00, 95% CI 2-sided [-2.00 to 0.00]

5. Secondary Outcome: Change From Baseline in the Investigator-Rated Conners' Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale (CAARS) Total Score at Week 2, Week 3, Week 4, and Week 5
Description: as for outcome 2
Time Frame: Baseline and Weeks 2, 3, 4, and 5
Population: Intent-to-Treat (ITT) Population (N), defined as subjects who were randomly assigned to one of two treatment groups, took at least 1 dose of study medication, and had a valid baseline CAARS assessment (pre-dosing) and at least one valid post-baseline CAARS assessment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IR Viloxazine | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale
  Raw Score; Baseline | 36.0 [20 to 54] | 35.0 [21 to 45]
  Change from Baseline score; Week 2 | -8.0 [-33 to 1] | -6.0 [-27 to 6]
  Change from Baseline score; Week 3 | -13.5 [-32 to -2] | -6.0 [-34 to 5]
  Change from Baseline score; Week 4 | -12.5 [-33 to -3] | -7.0 [-31 to 5]
  Change from Baseline score; Week 5 | -13.0 [-37 to 9] | -7.0 [-32 to 7]
Statistical Analysis 1: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 2 data; Test type: Superiority; p = 0.6022, Wilcoxon (Mann-Whitney); Median Difference (Net) = 1.00, 95% CI 2-sided [-4.00 to 6.00]
Statistical Analysis 2: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 3 data; Test type: Superiority; p = 0.0794, Wilcoxon (Mann-Whitney); Median Difference (Net) = -4.00, 95% CI 2-sided [-10.0 to 1.00]
Statistical Analysis 3: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 4 data; Test type: Superiority; p = 0.0747, Wilcoxon (Mann-Whitney); Median Difference (Net) = -6.00, 95% CI 2-sided [-10.0 to 0.00]
Statistical Analysis 4: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 5 data; Test type: Superiority; p = 0.0545, Wilcoxon (Mann-Whitney); Median Difference (Net) = -6.50, 95% CI 2-sided [-12.0 to 0.00]

6. Secondary Outcome: Change From Baseline in the Self-rated Conners' Adult Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale (CAARS) Total Score at Week 6
Description: as for outcome 2
Time Frame: Baseline and Week 6
Population: as for outcome 5
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IR Viloxazine | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale
  Raw score; Baseline | 35.0 [7 to 49] | 34.0 [13 to 48]
  Change from Baseline score; Week 6 | -10.5 [-46 to 7] | -1.0 [-35 to 8]
Statistical Analysis 1: Comparison: IR Viloxazine vs Placebo; This analysis applies to Week 6 data; Test type: Superiority; p = 0.0349, Wilcoxon (Mann-Whitney); Median Difference (Net) = 7.00, 95% CI 2-sided [1.00 to 13.00]

7. Secondary Outcome: Global Clinical Impression-Improvement (CGI-I) Score at Week 1, Week 2, Week 3, Week 4, Week 5, and Week 6
Description: The Global Clinical Impression-Improvement (CGI-I) scale is a single item clinician-rated assessment of how much the subject's condition (symptoms) has improved, worsened, or has not changed relative to his/her baseline state prior to the beginning of treatment; it is rated on a 7-point scale from 1 to 7, where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse. A CGI-I score <4 represents a better outcome.
Time Frame: Weeks 1, 2, 3, 4, 5, and 6
Population: Intent-to-Treat (ITT) Population (N), defined as subjects who were randomly assigned to one of two treatment groups, took at least 1 dose of study medication, and at least one valid post-baseline CGI-I assessment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | IR Viloxazine | Placebo
Number analyzed (Participants) | 26 | 25
units on a scale
  Week 1 | 5.0 [3 to 7] | 5.0 [3 to 6]
  Week 2 | 4.0 [3 to 6] | 5.0 [2 to 6]
  Week 3 | 3.5 [3 to 5] | 5.0 [2 to 6]
  Week 4 | 4.0 [2 to 5] | 5.0 [2 to 6]
  Week 5 | 4.0 [2 to 5] | 5.0 [2 to 6]
  Week 6 | 3.5 [2 to 5] | 5.0 [2 to 6]
Statistical Analysis 1: Comparison: IR Viloxazine vs Placebo; Analysis pertains to Week 1 data; Test type: Superiority; p = 0.4038, Wilcoxon rank-sum test; Median Difference (Net) = -0.50, 95% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 2: Comparison: IR Viloxazine vs Placebo; Analysis pertains to Week 2 data; Test type: Superiority; p = 0.4460, Wilcoxon rank-sum test; Median Difference (Net) = -0.50, 95% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 3: Comparison: IR Viloxazine vs Placebo; Analysis pertains to Week 3 data; Test type: Superiority; p = 0.0549, Wilcoxon rank-sum test; Median Difference (Net) = -0.50, 95% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 4: Comparison: IR Viloxazine vs Placebo; Analysis pertains to Week 4 data; Test type: Superiority; p = 0.0759, Wilcoxon rank-sum test; Median Difference (Net) = -0.50, 95% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 5: Comparison: IR Viloxazine vs Placebo; Analysis pertains to Week 5 data; Test type: Superiority; p = 0.0342, Wilcoxon rank-sum test; Median Difference (Net) = -0.50, 95% CI 2-sided [-1.00 to 0.00]
Statistical Analysis 6: Comparison: IR Viloxazine vs Placebo; Analysis pertains to Week 6 data; Test type: Superiority; p = 0.0474, Wilcoxon rank-sum test; Median Difference (Net) = -1.00

ADVERSE EVENTS:
Time Frame: Weeks 1-6 of Treatment
Description: Safety Population, defined as subjects who were randomly assigned to one of two treatment groups and took at least one dose of study medication
Arm/Group | IR Viloxazine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 23/26 | 18/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IR Viloxazine (N=26) | Placebo (N=25)
Dry eye (Eye disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 10 | 2
Fatigue (General disorders) | 3 | 1
Irritability (General disorders) | 3 | 1
Nasopharyngitis (Infections and infestations) | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Weight decreased (Investigations) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 8 | 1
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 8 | 9
Hypogeusia (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 3 | 2
Abnormal dreams (Psychiatric disorders) | 3 | 0
Initial insomnia (Psychiatric disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2010-06-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT01107496/Prot_000.pdf
  • Statistical Analysis Plan (2011-02-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT01107496/SAP_001.pdf